CLINICAL TRIAL: NCT04881344
Title: Mucopexy Versus Laser Hemorrhoidoplasty for the Treatment of Hemorrhoidal Disease, a Prospective Randomized Controlled Trial
Brief Title: Mucopexy Versus Laser Hemorrhoidoplasty for the Treatment of Hemorrhoidal Disease
Acronym: MuLa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ris Frederic (Other)
Responsible Party: Sponsor-Investigator, Ris Frederic, Clinical Professor Frédéric Ris, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01375
Record Dates: First submitted 2021-05-02; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The laser hemorrhoidoplasty (laser group, intervention group) (Experimental)
  Interventions: Procedure: laser hemorrhoidoplasty
- The hemorrhoidopexy (mucopexy group, control group) (Active Comparator)
  Interventions: Procedure: mucopexy

INTERVENTIONS:
Procedure: laser hemorrhoidoplasty — * Under local anesthetic (or general anesthetic if contraindications to local anesthetic),
  * A laser optic fiber connected to a diode platform (Leonardo, Biolitec AG, Jena, Germany) will be applied threw a anoscope. After making a 1-mm opening at the external border of hemorrhoid pocket, the fiber will be introduced in the hemorrhoidal tissue. Several pulses, each lasting for 1.2 s, with a 0.6-s pause between pulses, will be delivered to the tissue.
  * As a day-case procedure (or short-stay if medical or social factors precluded ambulatory intervention),
  * Postoperative care will consist of: normal diet, bulking laxatives, self-irrigation to the anal wound at six times per day and painkiller. Absence for work certificate will be made for 7 days for each patient and they will be told to return to work and normal daily activities as soon as they felt able.
  Arms: The laser hemorrhoidoplasty (laser group, intervention group)
Procedure: mucopexy — * Threw an anoscope, the hemorrhoidal cushion will be sutured using a half-circle (size 26) needle with a 2-0 poliglecaprone (Monocryl®, Ethicon, USA). Then, a continuous suture will be performed on the mucosa of the anal canal, and will terminate above the dentate line. The hemorrhoidal artery will be ligated by this suture. Then, the ligation will be tied to realize the hemorrhoidopexy.
  * Same anesthetic technique and postoperative care as the intervention group. As a day-case procedure (or short-stay if medical or social factors precluded ambulatory intervention).
  Arms: The hemorrhoidopexy (mucopexy group, control group)

SUMMARY:
Hemorrhoidal disease is a frequent anorectal disorder and the main reason for a visit to a coloproctologist. Hemorrhoids are present in healthy individuals. However, they can become pathologic, manifesting with pain, prolapse, itching, bleeding or soiling. Initially, they can be managed conservatively. When this failed to cure the symptoms, surgical therapy is indicated. For grade II (hemorrhoids prolapsing during straining but reducing spontaneously) or grade III (hemorrhoids prolapsing during straining but requiring manual reduction), laser hemorrhoidoplasty or mucopexy are safe and efficient procedures to treat hemorrhoids. However, the optimal treatment is still under debate. Recently, a randomized controlled trial reported lower recurrence and faster return to work associated with laser therapy. We aimed to compare both therapies, to assess the benefits of laser therapy for the treatment of hemorrhoidal disease symptoms, using a validated score.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Hemorrhoidal disease grade II to III unresponsive to medical therapy
* Age ≥18

Exclusion Criteria:

* Inability to follow the procedures of the study,
* Enrollment of the investigator, his/her family members, employees and other dependent persons,
* Anesthesiology contraindications to surgery,
* Emergency situation,
* Hemorrhoids associated with pregnancy,
* Oher surgical intervention performed at the same time of the hemorrhoids treatment,
* Concomitant anorectal disorders (fissure, fistula), thrombosed hemorrhoid,
* Previous pelvic radiotherapy, previous proctologic intervention during the last three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The Symptom Score | 6 postoperative months
  The primary outcome will be the "Symptom Score" at six postoperative months. This score ranges from 0 to 15 points, based on each of the five cardinal symptoms of hemorrhoidal disease (pain, itching, bleeding, discharge and prolapse) attributed from 0 to 3 points according to the frequency of their manifestation (0 point: never, 1 point: > 1x/month, <1x/week, 2 points: 1-6x/week, 3 points: 1x/day).

IPD SHARING:
Plan to Share IPD: No